CLINICAL TRIAL: NCT03427983
Title: Hydrodissection as a Treatment for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Peter C. Amadio, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-009840
Record Dates: First submitted 2018-01-25; First posted 2018-02-09 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized blinded study looking at two different ways of drug administration rather than the drug itself. We will compare ultrasound guided injection with hydrodissection to ultrasound guided injection without hydrodissection. In both groups, the active drug is the same in type and amount.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- US-guided regular injection (Other): US in-plane injection with corticosteroid and 1cc of lidocaine. Total of 2cc.
  Interventions: Procedure: Regular Injection
- US-guided hydrodissection (Other): US in-plane injection with corticosteroid and 1cc of lidocaine, and 3cc of saline. Total of 5cc.
  Interventions: Procedure: Hydrodissection

INTERVENTIONS:
Procedure: Hydrodissection — Additional 3cc's of saline is used to establish an increase in hydrodissection during routine treatment.
  Arms: US-guided hydrodissection
Procedure: Regular Injection — Corticosteroid and lidocaine injection without additional saline is used as routine treatment.
  Arms: US-guided regular injection

SUMMARY:
This is a pilot study designed to acquire data on the added value of hydrodissection when using a corticosteroid injection as a treatment for patients with carpal tunnel syndrome. Hydrodissection is part of a standard clinical care injection under ultrasound guidance in which the fluid is used to separate the nerve from surrounding structures.

ELIGIBILITY:
Inclusion Criteria:

* Clinical CTS diagnosis with indication for steroid injection as determined by attending physician (if both hands are involved, only the side with the most severe CTS as indicated by electromyography (EMG) will be included) AND
* adult men and women between age 21 and 80 AND
* no more than moderate severity as indicated by EMG AND
* symptoms of numbness or tingling for at least 4 weeks in the median nerve distribution area AND
* classic or probable carpal tunnel syndrome on Katz-Stirrat hand diagram AND
* ability to complete English-language questionnaires and clinical evaluations AND
* is reachable by phone for the follow up contact

Exclusion Criteria:

Exclusion criteria are largely based on the premises of only including patients with idiopathic carpal tunnel syndrome without expected interferences of the acquisition of the ultrasound images or corticosteroid treatment.

* Previous Carpal Tunnel Release (CTR) or other volar wrist surgery on the study hand OR known tumor/mass OR deformity of the study hand/wrist OR
* previous history of steroid injection into carpal tunnel OR
* currently taking a steroid medication either regularly or on an as needed basis OR
* any of the following clinical diagnoses or conditions: Cervical radiculopathy; rheumatoid or other inflammatory arthritis, including gout; osteoarthritis in the wrist; renal failure; sarcoidosis; peripheral nerve disease; diabetes, thyroid disease or other metabolic disorder; pregnancy; amyloidosis; or major trauma (fractures or complete ligamentous tears) to the ipsilateral arm OR
* prisoners, institutionalized individuals, or others who may be considered vulnerable populations, such as individuals with dementia

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Tolerance | 6 months
  Acquire data on the added value of hydrodissection when using injection as a treatment for patients with Carpal Tunnel Syndrome (CTS). Questionnaires will be used to assess level of tolerance using a 10 point Likert Scale.

SECONDARY OUTCOMES:
Clinical Severity of Carpal Tunnel Syndrome | 6 months
  The Boston Carpal Tunnel Assessment questionnaire will be used to assess both symptom severity and functional status using a 19 item questionnaire with scores between values 1-5.
Overall Pain | 6 months
  The visual analog scale will be used to assess overall pain. This is a 1-10 Likert scale.
Additional Treatment | 6 months
  After 6 months patients will be asked whether they have had additional treatment for their Carpal Tunnel Syndrome after the ultrasound guided injection. The date, location, and time frame of the additional treatment will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Amadio, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States